CLINICAL TRIAL: NCT06292455
Title: Association of Hand and Forearm Anthropometrics With Grip Strength and Forehand Smash Quality Following Six-week Elastic Resistance Training in Collegiate Badminton Players
Brief Title: Association of Anthropometrics With Grip Strength and Smash Quality Post Six Week Elastic Resistance Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RIPHAH/RCRS/REC/00713
Record Dates: First submitted 2020-11-15; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Anthropometric Measurements and Elastic Resistance Training; Sports Physical Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Elastic resistance training (Experimental): elastic resistance training of upper limb
  Interventions: Other: Elastic resistance training
- Conventional resistance training (Other): players follow their routine exercise protocol
  Interventions: Other: Conventional Resistance Training

INTERVENTIONS:
Other: Elastic resistance training — six-weeks elastic resistance training of upper limb. Three days per week. volume per session would be 10 repetitions and three sets. 2 minute rest interval between each set.
  Arms: Elastic resistance training
Other: Conventional Resistance Training — players follow their routine exercise protocol
  Arms: Conventional resistance training

SUMMARY:
To determine the association of hand and forearm anthropometrics on grip strength and forehand smash quality of badminton players after six-weeks of elastic resistance training.

DETAILED DESCRIPTION:
As literature suggests that anthropometrics such as BMI and height do affect many game outcomes but specific anthropometrics have not been considered before so it is included in this study. Similarly the affects of elastic resistance training for lower limb has been recorded while the literature lacks for upper limb.

ELIGIBILITY:
Inclusion Criteria:

* collegiate players of Badminton.
* Players attending at least two training sessions per week for the past one month

Exclusion Criteria:

* Players having strain or sprain of upper or lower limb within the last months
* Payers having any cardiovascular, neuromusculoskeletal or other systematic pathology.

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2020-07-10 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Smash quality (Power) | BAseline to six-week
  Power is measured in watts
Smash quality (Speed) | BAseline to six-week
  Measured in meter per second
Smash quality (Distance) | BAseline to six-week
  Measured in meter

CONTACTS AND LOCATIONS:
Overall Officials: Waqar Ahmad Awan, Phd, Principal Investigator — Riphah International University
Locations (1):
- Riphah international University, Islamabad, ICT, Pakistan

IPD SHARING:
Plan to Share IPD: No